CLINICAL TRIAL: NCT04099108
Title: The Effect of Combined Intravenous, Bolus Amino Acid Supplementation and Mobilisation on Skeletal Muscle During the Acute Phase of Critical Illness: a Randomised Controlled Trial.
Brief Title: Effect of Combined IV Bolus Amino Acid Supplementation and Mobilisation on Skeletal Muscle During the First 10 Days in the ICU: A RCT
Acronym: ProMob-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: Fresenius Kabi (Industry); University of the Western Cape (Other)
Responsible Party: Principal Investigator, Prof Renee Blaauw, Professor, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VAMI-001-IP4; VAMI-001-IP4 (Other Grant/Funding Number: Fresenius Kabi JUMPStart Research Grant)
Record Dates: First submitted 2019-09-18; First posted 2019-09-23 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2022-01

CONDITIONS: Critical Illness
Keywords: critical illness, amino acids, mobilisation, muscle
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Owing to the nature of the intervention, blinding of participants and treating clinicians was not feasible. However, blinding was maintained for primary outcome assessments, namely: (1) laboratory personnel responsible for biopsy analyses were blinded to group allocation, and (2) ultrasound image analysis was conducted by a blinded assessor. Furthermore, investigators responsible for secondary outcome measures with a subjective component, i.e., MRC sum score and 6MWT assessment, were blinded. Recognising the importance of clearly reporting blinding procedures in RCTs to enhance internal validity and adhere to CONSORT recommendations, the following measures were implemented:
  * The combined study intervention was performed in the morning, and outcome assessments were blinded in the afternoon with a sufficient interval to avoid overlapping.
  * The participants were prompted not to disclose their perceptions of group allocation during the outcome assessments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Combined cycle ergometry and bolus amino acid supplementation, along with standard of care
  Interventions: Combination Product: Combined cycle ergometry and bolus amino acid supplementation
- Control (No Intervention): Standard of care only (standard care nutrition guided by the ESPEN 2019 guidelines, and routine mobilisation performed as per the local unit's protocols and practice)

INTERVENTIONS:
Combination Product: Combined cycle ergometry and bolus amino acid supplementation — A 4-hour intravenous amino acid bolus combined with 45 minutes of cycle ergometry initiated within 1 hour of initiation of the amino acid supplement, starting on ICU Day 3-4 and given daily for a minimum of 5 days, and until latest Day 10 in the ICU.
  Arms: Intervention

SUMMARY:
A single-centre, two-arm, parallel randomised controlled trial (RCT) to compare the combined effect of early intravenous bolus amino acid supplementation and mobilisation versus standard of care on changes in muscle mass over the first week in ICU. Half of study participants will receive the study intervention (an intravenous bolus amino acid supplement combined with in-bed cycling), while the other half will receive standard of care only.

DETAILED DESCRIPTION:
Critical illness survivors often suffer from severe muscle mass depletion and a profound long-term functional impairment. Hence effective strategies, or a combination of strategies, are needed to reduce skeletal muscle wasting during critical illness. Although amino acids and mobilisation are both known to stimulate the mechanistic target of rapamycin pathway (MTOR) pathway for muscle protein synthesis in healthy adults, there are no trials to date investigating the combined approach of combined cycle ergometry and bolus amino acid supplementation on muscle accretion in the ICU.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years) admitted to medical/surgical ICU of Tygerberg Academic Hospital (TBH)
* Expected length of mechanical- or non-invasive ventilation > 48 hours
* Receiving enteral (EN) and/or parenteral nutrition (PN) as per standard care and for a minimum of 5 days
* Expected ICU length of stay of 7 days

Exclusion Criteria:

* Spinal cord lesion or intracranial process associated with muscle weakness
* Acute/chronic degenerative neuromuscular condition
* Fulminant hepatic failure/severe chronic liver disease (MELD score ≥20) or renal failure (based on KDIGO) not on Renal Replacement Therapy
* Untreated thrombosis, or thrombosis where therapeutic levels of anticoagulants have not been reached at the time of inclusion
* Any condition deemed inappropriate by the overseeing doctor- such as precautions or contraindications related to the movement as a result of trauma and/or surgery to the spine, pelvis or lower limbs, or haemodynamic instability.
* Other: imminent death or withdrawal of treatment, pregnancy, lower limb amputation/s or fractures, readmission after previous randomisation, long-term corticosteroid therapy, morbidly obese (BMI ≥ 40kg/m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in vastus lateralis myofiber cross-sectional area (biopsy) from pre- to post-intervention. | Pre-intervention biopsy performed 1 day before initiating the combined study intervention (on average day 2). Post-intervention biopsy performed after completing 5-days of the combined study intervention (on average day 8).
Change in rectus femoris muscle cross-sectional area (ultrasound) from pre- to post-intervention | Pre-intervention biopsy performed 1 day before initiating the combined study intervention (on average day 2). Post-intervention biopsy performed after completing 5-days of the combined study intervention (on average day 8).

SECONDARY OUTCOMES:
Change in protein-to-DNA ratio as a secondary marker of muscle mass | From pre- to post-intervention
  Obtained from muscle biopsy of the musculus vastus lateralis of the quadriceps
Signalling pathways for muscle protein synthesis and breakdown | From pre- to post-intervention
  Key proteins regulating muscle protein synthesis and breakdown, including markers of autophagy
Change in muscle mass (rectus femoris muscle CSA) and quality (RF muscle echogenicity) over shorter intervals from pre-intervention until study exit (Pre-intervention, Day 5, 7, 10, study exit) | Over shorter intervals from pre-intervention until study exit, if possible (Pre-intervention, Day 5, 7, 10, study exit)
Change in plasma amino acid levels (intervention group only) | Plasma samples will be obtained at 3 time intervals, (1) prior to amino acid infusion (T0), (2) 4 hours post amino acid infusion (T1), and (3) 24 hours post amino acid infusion (T2)
  Based on plasma samples obtained on ICU day 5
Muscle strength | Performed upon ICU awakening, and repeated on ICU discharge and study exit (day 28 or hospital discharge if earlier)
  Overall muscle strength will be evaluated using the Medical Research Council (MRC) sum-score via standardised "manual muscle testing" with each of 12 muscle groups assessed using a 6-point MRC scale and summed to a total score (range: 0 - 60)
Physical capability | Performed on study exit only (day 28, or day of hospital discharge if discharged earlier)
  Based on 6-minute walking test

OTHER OUTCOMES:
Change in measured energy expenditure over the first 10 days in ICU | From ICU Day 3+-1 until ICU Day 10+-1, unless contraindicated.
  Indirect calorimetry measurements performed as part of standard care nutrition on alternate days from ICU Day 3+-1 until ICU Day 10+-1 in all participants, unless contraindicated, were analysed to assess the change in MEE over time (across the cohort)
Assess phase angle (from BIA) as a potential surrogate marker of muscle mass & quality. | Pre- and post-intervention timepoints
  Assess correlation between whole-body phase angle and vastus lateralis myofiber CSA (biopsy), rectus femoris muscle CSA (ultrasound) and rectus femoris echogenicity.
Change in Urea-to-Creatinine Ratio (UCR) over the first 10 days of ICU admission and its correlation with markers of muscle mass | Over first 10 days of ICU admission
  To investigate the effect of the combined intervention, compared with standard care alone, on the change in Urea-to-Creatinine Ratio (UCR) over the first 10 days of ICU admission and to assess the correlation between UCR and biopsy myofiber CSA and ultrasound muscle CSA as markers of muscle mass.

CONTACTS AND LOCATIONS:
Overall Officials: Lizl Veldsman, M Nutr, Principal Investigator — University of Stellenbosch
Locations (1):
- Tygerberg Hospital, Cape Town, Western Cape, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Veldsman L, Lupton-Smith A, Richards GA, Blaauw R: Muscle ultrasound: a reliable bedside tool for dietitians to monitor muscle mass, South Afr J Clin Nutr. 2024:37(3): 125 - 130. doi: 10.1080/16070658.2024.2363707.
- [Result] Veldsman L, Richards GA, Lombard C, Blaauw R. Course of measured energy expenditure over the first 10 days of critical illness: A nested prospective study in an adult surgical ICU. Clin Nutr ESPEN. 2025 Feb;65:227-235. doi: 10.1016/j.clnesp.2024.11.009. Epub 2024 Nov 16. PMID 39551349